CLINICAL TRIAL: NCT06205953
Title: Bonding Molecular Genotyping and Phenotyping to Outcome Measures in AL Amyloidosis: A EUropean REgistry and Sample Sharing networK to Promote the Diagnosis and Management of Light Chain Amyloidosis (EUREKA)
Brief Title: A EUropean REgistry and Sample Sharing networK to Promote the Diagnosis and Management of Light Chain Amyloidosis (EUREKA)
Acronym: EUREKA
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giovanni Palladini, MD, PhD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: AC-021-EU
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood, bone marrow aspirate, serum, plasma, urine, fat tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective patients' registry collecting all new cases of AL amyloidosis evaluated at referral Centers from across Europe and a sample sharing network will be created to study mechanisms of the disease through the use of advanced molecular technologies and big data analysis tools.

DETAILED DESCRIPTION:
In the frame of the EUREKA Consortium, a patients' registry collecting all new cases of AL amyloidosis evaluated at referral Centers across Europe or at their satellite sites will be created, in association with a cross-border biorepository and sample sharing network for the study of both disease-causing light chains and plasma cells with advanced molecular technologies. A dedicated site will support the Consortium with big data analysis and artificial intelligence applied to health. The aims are: 1) Defining the impact of advanced molecular technologies to promote early diagnosis and guide therapeutic choices; 2) describing the natural history of the disease in a representative cohort of AL patients in the contemporary era of effective anti-plasma cell therapies; 3) investigating and refining novel advanced technologies to detect with high sensitivity residual disease-causing plasma cells/light chains in patients achieving a complete hematologic response to therapy (minimal residual disease, MRD).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of systemic AL amyloidosis;
* treatment-naïve;
* age ≥18 years;
* ability to understand and willingness to sign an informed consent;
* planned follow-up at participating center.

Exclusion Criteria:

* non-AL amyloidosis;
* previous treatment for AL amyloidosis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 patients with AL amyloidosis will be enrolled at diagnosis and evaluated at any of the participating clinical centers.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality at 24 months by stage | 24 months from diagnosis
  Mortality at 24 months by stage will be evaluated

SECONDARY OUTCOMES:
Rate of hematologic relapse in Complete Response patients at 2 years by MRD status | 2 years from diagnosis
  Rate of hematologic relapse in Complete Response patients at 2 years by MRD status will be evaluated

CONTACTS AND LOCATIONS:
Locations (6):
- Medical Department, Amyloidosis Center, University Hospital, Im Neuenheimer Feld 672, Heidelberg, Germany
- Fondazione IRCCS Policlinico San Matteo, Pavia, Viale Golgi 19, 27100, Pavia, Italy
- UMC Utrecht, dept Hematology, Amyloid Expertise Center, Utrecht, Heidelberglaan, Utrecht, Netherlands
- Instituto de Investigación Sanitaria de Navarra (IdiSNA) C. de Irunlarrea, 3, 31008 Pamplona, Navarra, Pamplona, Spain
- University of Applied Sciences and Arts Northwestern Switzerland, Institute of Medical Engineering and Medical Informatics, Muttenz, Switzerland
- Universidad de la Republica Hospital de Clinicas "Dr Manuel Quintela", Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No